CLINICAL TRIAL: NCT00918047
Title: Multiple Dose, Open-Label, Multi-Center Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of OXC XR as Adjunctive Therapy in Pediatric Subjects With Refractory Partial Epilepsy
Brief Title: Study of PK and Safety of OXC (Oxcarbazepine) XR (Extended Release) as Adjunctive Therapy in Pediatric Epilepsy Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 804P107
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Epilepsies, Partial
MeSH Terms: conditions — Epilepsies, Partial | interventions — Oxcarbazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- SPN-804O 150mg/Day (Experimental): Subjects who weighed 15.0 to 29.9 kg dosed with SPN-804O 150mg/Day
  Interventions: Drug: SPN-804O
- SPN-8040 300mg/Day (Experimental): Subjects who weighed 30.0 to 44.9 kg dosed with SPN-8040 300mg/Day
  Interventions: Drug: SPN-804O
- SPN-8040 450mg/Day (Experimental): Subjects who weighed 45.0 to 59.9 kg dosed with SPN-8040 450mg/Day
  Interventions: Drug: SPN-804O
- SPN-8040 600mg/Day (Experimental): Subjects who weighed 60.0 kg and above dosed with SPN-8040 600mg/Day
  Interventions: Drug: SPN-804O

INTERVENTIONS:
Drug: SPN-804O — Open Label study
  Other Names: oxcarbazepine extended-release; OXC XR; Oxtellar XR

SUMMARY:
Study to evaluate the pharmacokinetics, safety, and tolerability of OXC XR as adjunctive therapy in pediatric subjects with refractory partial epilepsy.

DETAILED DESCRIPTION:
This was an open-label, multiple dose, multicenter study consisting of a Screening Period (up to 14 days), a Dosing Period (7 days), and a Follow-up Period (7 days). In-clinic visits occurred at screening, Visit 1 (Day 0), and Visit 2 (Day 7)/Early Discontinuation. All subjects received open-label SPN 804O as adjunctive therapy during the Dosing Period. At Visit 1, eligible subjects were assigned to 1 of 4 treatment groups (150, 300, 450, or 600mg/day) based on weight (15-<30, 30-<45, 45-<60, >=60kg). The Dosing Period consisted of six consecutive days of a daily dose, taken at home, followed by a final day with the dose taken on-site and including blood draws for PK analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed assent (IAF), as appropriate, with written informed permission (and informed consent (ICF) where required by regional laws or regulations) from the parent or legally-authorized representative (LAR).
2. Male or female aged 4 to 17 years, inclusive, with a current diagnosis of partial onset seizures with or without secondarily generalized seizures as confirmed by the 1981 and 1989 International League Against Epilepsy Classifications).
3. Currently receiving treatment with at least one and up to two anti-epileptic drugs (AEDs), excluding oxcarbazepine and phenytoin. AED therapy must have been initiated more than one month prior to Visit 1 and doses must be stable for at least two weeks prior to Visit 1. A vagal nerve stimulator implanted for at least six months and with parameters unchanged for at least one month prior to Visit 1 is allowed and not considered to be an AED. Magnet use is allowed.
4. No diagnosis of a progressive neurological disorder based on previous imaging.
5. Weight within the 25 - 75 % weight-for-age percentiles based on the National Center for Health Statistics Growth Charts, and not less than 15.0kg.
6. Able and willing to swallow whole tablets.
7. Females of childbearing potential (FOCP) should either be sexually inactive (abstinent) for 14 days prior to the first dose, throughout the study and for four days following the last dose or, if sexually active, will be using one of the following acceptable birth control methods:

   1. Surgically sterile (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) six months minimum;
   2. Intrauterine device in place for at least three months;
   3. Barrier methods (condom, diaphragm) with spermicide for at least 14 days prior to the first dose, throughout the study and for four days following the last dose;
   4. Surgical sterilization of the partner (vasectomy for six months minimum);
   5. Hormonal contraceptives in addition to a barrier method (condom, diaphragm) with spermicide for at least 14 days prior to the first dose, throughout the study and for four days following the last dose.

Exclusion Criteria:

1. A documented history of status epilepticus in the past year.
2. Seizures secondary to illicit drug or alcohol use, infection, neoplasia, demyelinating disease, degenerative neurological disease, or central nervous system disease deemed progressive, metabolic illness, or progressive degenerative disease.
3. Diagnosis or an electroencephalogram consistent with a diagnosis of seizure disorders other than partial epilepsy.
4. Meets criteria for history of major depressive or manic episode, according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition Text Revision.
5. Any history of suicide intent and/or attempt.
6. History or presence of clinically significant, chronic medical condition, especially those contraindicating antiseizure medication, (e.g., any neurological, gastrointestinal, endocrine, cardiovascular, pulmonary, hematological, immunologic, renal, hepatic or metabolic disease) that may affect the safety of the subject in the opinion of the Investigator.
7. Use of oxcarbazepine or phenytoin within 10 days prior to first dose of SM.
8. Use of felbamate with less than 18 months of continuous exposure prior to screening.
9. Frequent need of rescue benzodiazepines (more than once in a 28 day period).
10. Use of diuretics or other sodium-lowering medications within seven days prior to first dose of study medication (SM).
11. History or presence of clinically significant laboratory, electrocardiogram (ECG), or vital sign abnormalities at screening that may affect the safety of the subject, in the opinion of the Investigator.
12. Presence of potential hepatic function impairment as shown by, but not limited to, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 times the upper limit of normal (ULN), or total bilirubin >1.5 times ULN.
13. Presence of suspected impairment of renal function defined by serum creatinine ≥1.5 times ULN.
14. History of substance abuse or dependence.
15. Females who are pregnant or lactating.
16. Previous known hypersensitivity to OXC or other related drugs, such as carbamazepine.
17. Use of an investigational drug or device or participation in an investigational study within 30 days prior to the first dose of SM.
18. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Examine the steady-state pharmacokinetics (PK) of OXC XR and to assess the safety and tolerability of repeated oral dosing of OXC XR in pediatric subjects with partial seizures.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Little Rock, Arkansas
  - Loxahatchee Groves, Florida
  - Tampa, Florida
  - Rockville, Maryland
  - Lake Success, New York
  - Rochester, New York
  - Kingsport, Tennessee
  - San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No